CLINICAL TRIAL: NCT06270342
Title: The Effect of Dual Task On Upper Extremity Functions In Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Eda Ozge OKUR, Asst. Prof., Kutahya Health Sciences University
Other Study IDs: DTMS
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: Dual Task; Dual Task Effect; Multiple Sclerosis; Upper Extremity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS: patients with multiple sclerosis
  Interventions: Other: dual task assessment
- Control: healthy volunteers
  Interventions: Other: dual task assessment

INTERVENTIONS:
Other: dual task assessment — The Minnesota Manual Dexterity Test was used to evaluate the upper extremity function of the participants in single and dual task conditions, and the Dual Task Questionnaire was used to evaluate the difficulties experienced during dual tasks. In the dual-task turning test, in addition to the single-task turning test, they were given a cognitive task, the task of counting the months of the year backwards from December to January. The dual-task turning test was continued by changing hands at the end of each turn until the last disk was turned. Meanwhile, verbal fluency and hand errors made while spinning the disc were recorded.

SUMMARY:
The primary aim of this study was to investigate the effect of dual tasking on upper extremity functions in individuals with multiple sclerosis (MS) and compare with healthy controls. Additionally, another aim of our study was to compare the cognitive status, quality of life, fatigue and emotional states of individuals with MS and healthy controls.

DETAILED DESCRIPTION:
The study was carried out at Kutahya Health Sciences University Evliya Çelebi Training and Research Hospital. 30 individuals with MS and 30 healthy controls, aged 18-65, were included in the study. In the evaluation, demographic and clinical data were recorded first. The Minnesota Manual Dexterity Test was used to evaluate the upper extremity function of the participants in single and dual task conditions, and the Dual Task Questionnaire was used to evaluate the difficulties experienced during dual tasks.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Multiple Sclerosis for at least 1 year
* Being between the ages of 18-65
* Being at least a primary school graduate
* Volunteering to participate in the study
* EDSS score between 1 and 6.5

Exclusion Criteria:

* Patients whose Multiple Sclerosis diagnosis is uncertain
* Having additional neurological disease that may affect clinical evaluation
* Having a neurological and/or psychiatric disease that may affect cognitive tests
* Having had an attack in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having been diagnosed with MS and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The Minnesota Manual Dexterity Test | 30 minutes
  Upper Extremity Function Evaluation. The Minnesota Manual Dexterity Test basically consists of two subtests, the placement and translation test.
  Completing the test faster indicates better dexterity.
Dual Task Questionnaire | 10 minutes
  Dual Task Difficulty Evaluation. The survey consists of 10 items and is scored out of 5 points per question.
  A higher total score indicates worse dual task performance.
Edinburgh Handedness Questionnaire | 10 minutes
  Hand Preference Evaluation. The total scoring is between 100 and -100, individuals with more than 40 points are given right hand; Individuals in this score range from 40 to -40 inclusive are recorded as those who use both hands actively, and individuals with scores of -40 points and below are recorded as left-handed.
Expanded Disability Status Scale | 10 minutes
  Disability Status Evaluation. A score of 0 on the scale indicates normal neurological status, while a score of 10 means MS-related death.
Brief International Cognitive Assessment Battery for Multiple Sclerosis | 15 minutes
  Cognitive Status Evaluation. BICAMS comprises three tests, the Symbol Digit Modalities Test (SDMT), the learning trials of the California Verbal Learning Test II (CVLT-II), and the Brief Visuospatial Memory Test-Revised (BVMT-R).
Beck Depression Scale | 10 minutes
  Emotional Status Evaluation. The lowest score that can be obtained from the scale is 0 and the highest score is 63. According to the resulting total score; It results in absence-mild, mild-moderate, moderate-severe or severe.
Fatigue Impact Scale | 5 minutes
  Fatigue Status Evaluation. Each question receives a score between 0 (no problem) and 4 (maximum problem). The highest score is 160, and higher scores indicate fatigue.
Multiple Sclerosis Quality of Life Questionnaire-54 | 15 minutes
  Quality of Life Status Evaluation. The survey contains 54 questions consisting of 12 sections. Added 18 questions are about; general quality of life (2 items), health stress (4 items), sexual functions and satisfaction (5 items), cognitive functions (4 items), energy (1 item), pain (1 item) and social functions (1 item).

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.